CLINICAL TRIAL: NCT01049542
Title: Effects of Urocortins on Forearm Arterial Blood Flow in Healthy Volunteers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Edinburgh (Other)
Responsible Party: Prof D E Newby, University of Edinburgh
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Basic Science
Other Study IDs: SV.Protocol1
Record Dates: First submitted 2010-01-12; First posted 2010-01-14 (Estimated); Last update posted 2010-11-16 (Estimated); Status verified 2010-11

CONDITIONS: Vascular Disease; Heart Disease
Keywords: Astressin 2B; Forearm blood flow; vascular; plethysmography; heart failure
MeSH Terms: conditions — Vascular Diseases; Heart Diseases; Heart Failure

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (1):
- Astressin 2B (Experimental): Healthy volunteers will receive incremental doses of intra arterial Astressin 2B (a selective and potent Urocortin 2 & 3 antagonist). This serves as a dose finding Protocol for Astressin 2B, which will be used in subsequent protocols.
  Interventions: Drug: Astressin 2B

INTERVENTIONS:
Drug: Astressin 2B — After an initial saline washout, increasing doses of Astressin 2B (at 0.032, 0.32, 3.2, 32, 320 and 3200 pmol/min) will be infused, for 10 minutes at each dose,intra arterially using forearm venous occlusion plethysmography. Forearm blood flow will be measured with each incremental dose of Astressin 2B.
  Other Names: Forearm vascular study

SUMMARY:
Impairment of the heart's pumping capacity (heart failure) remains a major clinical problem with a poor prognosis and the search for novel treatments remains an important area of research.

Urocortins are proteins that appear to increase blood flow and heart pumping activity. There has been particular interest in the role of Urocortins 2 & 3 (subtypes of Urocortins) in heart failure.

In this study, we will examine the effects and mechanisms of Urocortins 2 & 3 and the Corticotrophin Releasing Hormone Receptor Type 2 (CRH-R2) receptor (through which urocortins act) on forearm blood flow and release of natural blood clot dissolving factors in the forearm circulation of healthy volunteers.

In this study, we will look at the role of the lining of the blood vessel (endothelium) in response to urocortin types 2 and 3. We hypothesise that urocortins 2 & 3 act via the endothelium to cause dilatation of the blood vessels and release of tissue-plasminogen activating factor (blood clot dissolving factor). We also hypothesise that urocortins have a role in maintaining the normal baseline level of blood flow in forearm arteries. In addition to the above, we will also look at the effect of temporarily blocking the effect of urocortins, using a specially designed blocker drug (Astressin 2B).

Utilising the well-established technique of 'forearm venous occlusion plethysmography', we will be able to focus on the local effects of urocortins on arterial blood flow in forearm vessels, without affecting this system in the body as a whole.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers between 18 - 65 years (inclusive)

Exclusion Criteria:

* Lack of informed consent
* Age <18 years > 65 years
* Current involvement in a clinical trial
* Severe or significant co-morbidity including bleeding diathesis, renal or hepatic failure
* Smoker
* History of anaemia
* Recent infective/inflammatory condition
* Recent blood donation (prior 3 months)
* Positive baseline urine test for drugs of abuse (including cannabinoids, benzodiazepines, opiates, cocaine and amphetamines)

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2010-05; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Change in forearm blood flow | 3 hours
  Absolute change in forearm blood flow with respect to baseline forearm blood flow resulting from infusion of the study drugs, using forearm venous occlusion plethysmography

SECONDARY OUTCOMES:
Principle safety assessment, heart rate and blood pressure | 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: David E Newby, PhD FRCP, Principal Investigator — University of Edinburgh
Locations (1):
- Wellcome Trust Clinical Research Facility, Royal Infirmary of Edinburgh, Edinburgh, Mid Lothian, United Kingdom